CLINICAL TRIAL: NCT04133363
Title: Clinical, Radiographic, and Histomorphometric Outcomes Following Ridge Preservation Using Leukocyte Platelet Rich Fibrin (L-PRF) and Freeze-Dried Bone Allograft (FDBA) Layered Technique: A Prospective, Randomized Clinical Trial
Brief Title: To Compare Ridge Preservation Technique Using Leukocyte Platelet Rich Fibrin (L-PRF) and Freeze-dried Bone Allograft (FDBA) Layered Technique vs L-PRF/FDBA and L-PRF Alone in Influencing Quantity and Quality of New Bone Formation in Grafted Extraction Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicolaas C. Geurs, DDS, MS, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300004112
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Ridge Preservation
Keywords: L-PRF; Bone Allograft; Ridge Preservation; Socket grafting; Bone regeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ridge preservation using L-PRF/ FDBA Layered (Experimental): Atraumatic tooth extraction following by socket grafting using L-PRF/FDBA layered technique
  Interventions: Procedure: Ridge preservation using L-PRF/FDBA layered technique
- Ridge preservation using L-PRF/ FDBA (Experimental): Atraumatic tooth extraction following by socket grafting using L-PRF/FDBA
  Interventions: Procedure: Ridge preservation using L-PRF/FDBA
- Ridge preservation using L-PRF (Experimental): Atraumatic tooth extraction following by socket grafting using L-PRF alone
  Interventions: Procedure: Ridge preservation using L-PRF

INTERVENTIONS:
Procedure: Ridge preservation using L-PRF/FDBA layered technique — Atraumatic tooth extraction following by socket grafting using L-PRF/FDBA layered technique
  Arms: Ridge preservation using L-PRF/ FDBA Layered
Procedure: Ridge preservation using L-PRF/FDBA — Atraumatic tooth extraction following by socket grafting using L-PRF/FDBA
  Arms: Ridge preservation using L-PRF/ FDBA
Procedure: Ridge preservation using L-PRF — Atraumatic tooth extraction following by socket grafting using L-PRF
  Arms: Ridge preservation using L-PRF

SUMMARY:
This study will evaluate the effect of Leukocyte Platelet Rich Fibrin and freeze-dried bone allograft in a layered technique on the bone quantity and quality following socket grafting in preparation for endosseous implant placement.

Pre (baseline)- and post-grafting (3 months) clinical as well as 2- and 3-dimensional radiographic measurements will be used to evaluate the dimensional ridge changes between sites grafted with L-PRF/FDBA layered technique vs. L-PRF/FDBA and L-PRF alone.

Histological analysis will be performed by a bone biopsy taken at time of surgical re-entry (after 3 months) of grafted sites to place the dental implant and assessed for differences in new bone formation between the three types of graft.

DETAILED DESCRIPTION:
This study is a prospective, three-arm randomized trial that will evaluate and compare the bone healing following ridge preservation of extraction sockets using either L-PRF/FDBA layered technique or L-PRF/FDBA or L-PRF alone in a total of 30 patients (10 in each arm).

Qualifying participants and defects will be randomized following a computerized permutation block to receive either technique on day of surgery. Tooth extraction will be performed with a flapless minimally invasive technique, followed by socket grafting with a randomized graft.

The mineralized cortico-cancellous bone allograft that will be used in this study will be obtained from the same donor, lot and tissue bank to account for variation in age, race, gender and related healing potential of different graft sources.

Bone core biopsies will be harvested at time of implant placement 3 months following socket grafting. Bone cores will then undergo histological and histomorphometrical analyses to determine qualitative and quantitative healing differences between three treatment groups.

Clinical measurements are gathered at 2 time points (grating and implant placement) at all defects and will be compared for differences.

Cone beam computed tomography (CBCT) initial scans are conducted immediately following socket grafting and second scans obtained prior to implant placement. Virtual implant planning software will be utilized to assess and compare the 2- and 3-dimensional changes for all defects.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and able to read and understand English informed consent document
* At least 18 years old.
* Must be a patient at the UAB School of Dentistry
* Patient is willing and able to comply with all steps of the study
* Hopeless single-rooted tooth planned to be replaced with a dental implant and with healthy adjacent teeth not planned for extraction.

Exclusion Criteria:

* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Pregnant women
* Patient is a poor compliance risk (i.e., poor oral hygiene, history of alcohol or drug abuse)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ridge Preservation Using L-PRF/ FDBA Layered | Ridge Preservation Using L-PRF/ FDBA | Ridge Preservation Using L-PRF
Started | 10 | 10 | 10
Completed | 8 | 9 | 6
Not Completed | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridge Preservation Using L-PRF/ FDBA Layered | Ridge Preservation Using L-PRF/ FDBA | Ridge Preservation Using L-PRF | Total
Number analyzed (Participants) | 8 | 9 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 3 | 11
  >=65 years | 4 | 5 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 12
  Male | 5 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 8 | 9 | 4 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Measurements of Clinical Dimensional Changes at Alveolar Ridge 3 Months After Ridge Preservation Procedure Using L-PRF Alone, L-PRF/FDBA, and L-PRF/FDBA Layered Technique
Description: Compare quantitative clinical alveolar ridge dimensions (in mm) 3 months after ridge preservation between the three groups. Clinically we will measure the bone width of the ridge at time of extraction and after three months during the implant placement procedure. The dimensional changes will be calculated by subtracting the follow measurement from the initial measurement.
Time Frame: From baseline to 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ridge Preservation Using L-PRF/ FDBA Layered | Ridge Preservation Using L-PRF/ FDBA | Ridge Preservation Using L-PRF
Number analyzed (Participants) | 8 | 9 | 6
mm | 0.88 (1.55) | 0.78 (3.8) | 0.83 (2.8)

2. Primary Outcome: Measurements of the Radiographic Dimensional Changes at Alveolar Ridge 3 Months After Ridge Preservation Procedure Using L-PRF Alone, L-PRF/FDBA, and L-PRF/FDBA Layered Technique
Description: Compare quantitative radiographic alveolar ridge dimensions (in mm) 3 months after ridge preservation between the three groups using a CBCT scan. The bone width at the extraction site will be measured on the CBCT taken directly after the extraction. The same measurement will be taken at the 3 month follow up CBCT. The dimensional changes will be calculated by subtracting the follow measurement from the initial measurement.
Time Frame: From baseline to 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ridge Preservation Using L-PRF/ FDBA Layered | Ridge Preservation Using L-PRF/ FDBA | Ridge Preservation Using L-PRF
Number analyzed (Participants) | 8 | 9 | 6
mm | 1.03 (0.91) | 0.48 (1.93) | 0.9 (0.9)

3. Primary Outcome: Assessments of the Histology of the Bone Harvested at the 3 Month Visit.
Description: Measure quantitative histologic characteristics of new bone between the three groups after 3 months of ridge preservation by quantifying the distribution (in %) of new vital bone at the healed socket site. The quality of the bone created will analyzed using a descriptive analysis.
Time Frame: 3 months
Population: From the twenty-three(23) patients, histomorphometric analysis was performed on fifteen bone core biopsies obtained from the healed sockets (five in each group).
Measure: Mean (Standard Deviation); unit: in %
Arm/Group | Ridge Preservation Using L-PRF/ FDBA Layered | Ridge Preservation Using L-PRF/ FDBA | Ridge Preservation Using L-PRF
Number analyzed (Participants) | 5 | 5 | 5
in % | 52.15 (9.63) | 58.26 (2.84) | 38.59 (10.12)

ADVERSE EVENTS:
Time Frame: Baseline to 3 months
Arm/Group | Ridge Preservation Using L-PRF/ FDBA Layered | Ridge Preservation Using L-PRF/ FDBA | Ridge Preservation Using L-PRF
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT04133363/Prot_SAP_000.pdf